CLINICAL TRIAL: NCT00003072
Title: Amifostine (Ethyol) as a Protectant in Metastatic Ovarian and Non-Small Cell Lung Cancer in Paclitaxel/Carboplatin-Treated Patients: A Comparative Trial
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic Ovarian Cancer or Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Purpose: Supportive Care
Other Study IDs: CDR0000065752; UCSF-H57841348101A; ALZA-UCSF-H57841348101A; NCI-V97-1334
Record Dates: First submitted 1999-11-01; First posted 2004-09-06 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Lung Cancer; Neurotoxicity; Ovarian Cancer
Keywords: stage III non-small cell lung cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage IV non-small cell lung cancer; neurotoxicity
MeSH Terms: conditions — Lung Neoplasms; Neurotoxicity Syndromes; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial | interventions — Amifostine; Carboplatin; Paclitaxel

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving the drugs in different combinations may kill more tumor cells.

PURPOSE: Randomized phase II double-blinded trial to study the effectiveness of paclitaxel and carboplatin given with either amifostine or placebo in patients with metastatic stage III or stage IV ovarian cancer or metastatic stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether patients with metastatic ovarian and non-small cell lung cancer receiving carboplatin and paclitaxel have significantly fewer neuropathic events when treated with amifostine.

OUTLINE: This is a randomized, parallel group, double blind, controlled study. Patients are randomized to either the amifostine or control group. All patients receive intravenous paclitaxel over 3 hours, followed by carboplatin once every 3 weeks for 6 cycles. Patients who are randomized to the amifostine group receive intravenous amifostine administered as a 15 minute infusion 30 minutes prior to paclitaxel therapy. Patients randomized to the control group receive an intravenous placebo solution. Patients are discontinued from the study if they have disease progression or unacceptable toxic effects after 2 cycles of treatment. Patients are followed monthly for 8 months post treatment.

PROJECTED ACCRUAL: A total of 80 patients will be accrued (40 with advanced ovarian cancer and 40 with advanced non-small cell lung cancer) within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage III/IV ovarian or non-small cell lung cancer

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: ECOG 0-2 Life Expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 3.0 mg/dL Renal: Creatinine no greater than 2 mg/dL Other: Not pregnant or nursing No history of platinum, paclitaxel or amifostine hypersensitivity Prior myelosuppressive events allowed No clinically significant ascites

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy within 1 month of study Endocrine therapy: Not specified Radiotherapy: No prior radiation therapy within 1 month of study Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 1997-05; Primary Completion 1998-10 (Actual); Study Completion 1998-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Ignoffo, PharmD, Study Chair — University of California, San Francisco
Locations (4):
- United States (4):
  - Oncology Service of San Francisco General Hospital Medical Center, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - UCSF/Mt. Zion Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California